CLINICAL TRIAL: NCT00502502
Title: Feasibility Study of the Assessment of Symptom-Related Cytokines in Lung and GI Cancer Patients Undergoing Chemoradiation Therapy
Brief Title: Assessment of Symptom-Related Cytokines in Lung and Gastrointestinal (GI) Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANS02-495
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Anal Cancer; Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Lung Cancer
Keywords: Anal Cancer; Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Lung Cancer; Questionnaire; Survey; Chemoradiation Therapy; Symptoms; Cytokines
MeSH Terms: conditions — Anus Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected to study the levels of cytokines in your blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptom-Related Cytokines Questionnaire
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Weekly questionnaires lasting about 30 minutes.
  Other Names: Survey

SUMMARY:
Primary Objectives:

* To determine the feasibility of a study that would describe changes of certain circulating inflammatory cytokines (interleukin-1, 6, 8, 10, 12, and tumor necrosis factor-alpha [TNF] and symptoms related to chemoradiation therapy (pre-therapy, during therapy and up to 3 months post-therapy) among patients with lung, esophageal, gastric, colorectal and anal cancer.
* To determine the feasibility of studying neurocognitive function in patients with non-small cell lung cancer (NSCLC) at presentation and during chemoradiation therapy to determine the prevalence, severity, and pattern of cognitive symptoms.

DETAILED DESCRIPTION:
One of the ways to learn about the symptoms of chemoradiation therapy is by looking at how certain proteins called cytokines (found in the blood) change during therapy. Another way is to look at how thinking and memory may be changed because of treatment.

Before therapy starts, you will be asked to complete several questionnaires during a visit to the Radiation Oncology clinic at M. D. Anderson. These questionnaires measure physical and emotional symptoms. These questionnaires should take about 30 minutes to finish. Lung cancer patients will also complete some cognitive (mental) questionnaires. During this visit, the research nurse will teach you how to use the telephone system for measuring symptoms. You will tell the system the most convenient times for the telephone calls. The date of the call will be at the same or close to the date of your weekly clinic visit.

Before you begin your chemoradiation treatments, you will have a sample of blood drawn (around 2½ tablespoons). The sample of blood will be used to measure levels of cytokines in your blood pre treatment.

You will have about 2½ tablespoons of blood drawn again when you start chemoradiation, and then once a week while you are receiving treatment. These cytokines may be related to symptoms experienced while having treatment for cancer. These blood tests are being done to study the levels of cytokines in your blood during, and after treatment for cancer.

Symptoms will be monitored weekly using an interactive voice response telephone system. During chemoradiation, the automated telephone system will call you once a week to ask you to rate your symptoms and how much the symptoms interfere in your daily life. The information collected by these calls is only being used for this research study.

At the end of the chemoradiation, lung cancer patients will again be given questionnaires to measure cognitive symptoms.

For lung cancer patients who are post-chemotherapy, your symptoms will be monitored weekly for 3 months after therapy using the interactive voice response telephone system. For esophageal, gastric, colorectal, and anal patients who are post-therapy, your symptoms will be monitored weekly for 6 weeks after therapy using the interactive voice response telephone system. About 30 days after chemoradiation, you will have 2½ tablespoons of blood drawn at your regularly scheduled clinic visit. If you are not scheduled for a 3 month clinic visit, we will contact your local physician for blood lab results.

This is an investigational study. About 225 evaluable patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for chemoradiation therapy at MDACC.
2. Adults > 18 years of age.
3. Diagnosis of lung, esophageal, gastric, colorectal, or anal cancer.
4. English-speaking.
5. Lives in the United States.
6. Adequate vision and hearing to use the IVR system.
7. Provides written informed consent.

Exclusion Criteria:

1. Patients with a current diagnosis of psychosis or dementia.
2. Patients who are unable to complete the assessment measures or refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with lung, esophageal, gastric, colorectal or anal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2002-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Patient Symptom Assessment (Questionnaire) | Weekly for 1-3 months post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org